CLINICAL TRIAL: NCT06304480
Title: Effect of The Partial Substitution of Animal Protein by Soya-Based Fermented Product on Human Gut Microbiome and Clinical Health Markers
Brief Title: Effect of The Substitution of Animal Protein by Soya-Based Fermented Product on Human Gut Microbiome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Collaborators: AIT Austrian Institute of Technology GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AFCRO-179
Record Dates: First submitted 2024-02-21; First posted 2024-03-12 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Gut Microbiome
Keywords: Gut Microbiome; Microbiota; Plant protein; Soya protein

STUDY DESIGN:
Intervention Model Description: Randomised, open label, controlled, parallel study in healthy males and females.
Masking Description: Randomised, open label, controlled, parallel study in healthy males and females.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 100g fermented Tofu (Experimental): Participants will consume 100 g Miso fermented tofu per day which may be consumed any way i.e. fried, grilled, baked, etc to taste or prepared from the list of recipes provided.
  Interventions: Dietary Supplement: 100g fermented Tofu
- Control (No Intervention): Participants will consume their regular diet

INTERVENTIONS:
Dietary Supplement: 100g fermented Tofu — * Participants will consume 100 g Miso fermented tofu per day which may be consumed any way i.e. fried, grilled, baked, etc to taste or prepared from the list of recipes provided.
  * Participants will consume the first Study Product on the day of their Visit 3 (Day 0) and will consume their last Study Product the day prior to Visit 5 (Day 56).
  * Participants will be instructed to return any unused Study Product at Visit 5 (Day 56).
  Arms: 100g fermented Tofu

SUMMARY:
There is a growing understanding of the functioning and interconnectedness of microbiomes in the food system which offers great potential for enabling the development of new solutions contributing to achieving important food and nutrition goals including those requested by FOOD 2030. Of relevance in this regard is the provision of sustainable and healthy protein sources. Because of the obvious environmental and climate concerns associated with the production of animal-derived protein, a transition is needed to healthier and more environment-friendly diets, including a moderate-level consumption of red and processed meat and greater emphasis on plant-based foods.

As well as impact of meat production on the climate, it is well established that eating a diet rich in red meat promotes the growth of gut microbiome members that drive or exacerbate inflammation. Plant protein does not have these associations, and in fact it is often accompanied by fibre ingestion, which favours growth of health-promoting gut microbes. Replacing meat with plant protein offers the prospect of improving consumer health by improving the gut microbiome. The EU funded project MICROBIOMES4SOY will assess the effect of replacing animal protein with soya-derived protein on the human gut microbiome and whether this replacement can reduce the risk of inflammation-related diseases by gut microbiome modulation. This knowledge will provide a baseline for establishing new dietary pathways making use of soya protein and support dietary transition for EU citizens.

DETAILED DESCRIPTION:
Randomised, open label, controlled, parallel study in healthy males and females.

* Screening/Run-in: 21 days
* Intervention phase: 56 days
* Follow-up phase: 14 days
* Total time: 91 days

At Visit 1 (Screening visit) Participants will attend the study site and the following procedures will be carried out:

* Participants will receive oral and written information about the study and be allowed to ask questions.
* Participants will sign the informed consent document.
* Inclusion and exclusion criteria will be reviewed.
* Demographic, health, and lifestyle data will be collected.
* Medical history will be collected.
* Prior concomitant medication will be recorded.
* Height and weight will be measured, and BMI calculated.
* Vitals (blood pressure, heart rate and temperature) will be recorded.
* Participant contraception method will be confirmed.
* A blood sample (14 mL) will be collected for safety analysis.
* For individuals of childbearing potential, a urine sample will be collected, and pregnancy test performed (regardless of contraceptive use or relationship status).
* Participants will be provided with a stool collection kit and instructions for collecting and storing. Participants will collect the stool sample at home, within 48 hours prior to the scheduled visit and bring it to the clinic.
* Participants will complete the food frequency questionnaire (FFQ).
* Participants will be provided with a 3-Day food diary and instructions on how to complete the document. Participants will return the completed diary at the next visit.

At Visit 2 Day -14, Participants will attend this study Visit and the following procedures will be carried out:

* Participants will return the collected stool sample and will be stored for further analysis.
* Participants will be provided with a urine collection kit and instructions for collecting and storing.
* Participants will be provided with a stool collection kit and instructions for collecting and storing. Participants will collect stool samples at home, within 48 hours prior to the scheduled visit and bring it to the clinic.

At Visit 3 Day 0, Participants will attend this study visit, having fasted overnight for at least 10-hours and the following procedures will be carried out:

* Participant's continued consent to study procedures will be confirmed.
* Inclusion/exclusion criteria will be reviewed.
* Concomitant medication/supplements will be recorded.
* Vitals (blood pressure, heart rate and temperature) will be recorded.
* A fasting blood sample (10 mL) will be collected for lipids and stored for biomarker analysis.
* For individuals of childbearing potential, a urine sample will be collected, and pregnancy test performed (regardless of contraceptive use or relationship status).
* Participants will return the collected stool samples and will be stored for further analysis.
* Participants will return the collected urine sample and will be stored for further analysis.
* Participant will return the 3-Day food diary.
* Participants will complete SF-36 RAND questionnaire.

Participants will be randomised into one of the two groups as follows,

* Arm 1: Intervention (replacing a portion of red meat with 100 g of fermented tofu)
* Arm 2: Control
* Participants will be supplied Study Product and instructions of dosing.
* Participants will be provided with a urine collection kit and instructions for collecting and storing.
* Participants will be provided with a stool collection kit and instructions for collecting and storing. Participants will collect stool samples at home, within 48 hours of the scheduled visit and bring them to the clinic.
* Participants will be provided with a 3-Day food diary and instructions on how to complete the document. Participants will return the completed diary at their next visit.
* Participants will be provided with dietary advice.

At Visit 4 (Remote) Day 28: Participants will be contacted remotely on day 28 and the following procedures will be carried out:

* Participant's continued consent to study procedures will be confirmed.
* Concomitant medication/supplements will be recorded.
* Adverse events will be recorded.
* Participants Study Product compliance will be assessed.

At Visit 5 Day 56, Participants will attend this study visit, having fasted overnight for at least 10-hours and the following procedures will be carried out:

* Participant's continued consent to study procedures will be confirmed.
* Concomitant medication/supplements will be recorded.
* Vitals (blood pressure, heart rate and temperature) will be recorded.
* Adverse events will be recorded.
* A fasting blood sample (10 mL) will be collected for lipids and stored for biomarker analysis.
* For individuals of childbearing potential, a urine sample will be collected, and pregnancy test performed (regardless of contraceptive use or relationship status).
* Participants will return the collected urine sample and will be stored for further analysis.
* Participants will return the collected stool samples and will be stored for further analysis.
* Participants will be provided with a stool collection kit and instructions for collecting and storing. Participants will collect the stool sample at home, within 48 hours of the scheduled visit and bring them to the clinic.
* Participant will return the 3-Day food diary.
* Participants will complete SF-36 RAND questionnaire.
* Participants will return any unused Study Product and compliance will be assessed.

Participants will return to the study site for Visit 6 (Follow-up Visit) at day 70, having completed the follow-up phase of the study. The following procedures will be carried out:

* Participant's continued consent to study procedures will be confirmed.
* Concomitant medication/supplements will be recorded.
* Adverse events will be recorded.
* Participants will return the collected stool sample and will be stored for further analysis.

Data processing & Management Data required for the analysis will be acquired and transferred electronically to a central database by means of an Electronic Data Capture system (the "EDC-tool"). The EDC-tool will comprise an eCRF, designed specifically for the present study. High security standards for the transfer and storage of study data are guaranteed using technologies such as encrypted data transfer, firewalls, and periodic backup to protect centrally stored data. The eCRF is based on the electronic data capture system developed by Clindox, which is fully compliant with and a Gold Member of the Clinical Data Interchange Standards Consortium. The eCRF will be hosted on a dedicated validated stand-alone server placed in a double locked server room. According to the standards of the data protection law, all data obtained in the course of the study will be treated with discretion in order to guarantee the rights of the Participant's privacy.

Monitoring The responsible monitor will contact and visit the clinical site regularly and will be allowed, on request, to review the various records of the study (CRFs/eCRFs and other pertinent data) provided that Participant confidentiality is maintained in accordance with local requirements and as specified in the contract. The monitor will review the study documents (e.g., CRFs) at regular intervals throughout the study, to verify the adherence to the protocol and the legibility, completeness, consistency, and accuracy of the data being entered on them. The monitor will have access to laboratory test reports and other Participant records needed to verify the entries on the CRF/eCRF. This source data verification may be carried out remotely.

Quality assurance and quality control All Study Product used will be subjected to quality control. Quality assurance audits will be performed by the Sponsor (or any health authority) during the course of the clinical study or after its completion.

Adverse Events (AE):

For purposes of this study all AEs reported will be unexpected. The causality assessment of an AE to the investigational and/or study procedure(s) product will be rated as Unrelated, Unlikely, Possible, Probable or Definite using accepted criteria for clinical trials. The severity of AEs will be recorded, including the start and stop dates for each change in severity, and graded on a five-point-scale in accordance with the Common Terminology Criteria for Adverse Events. The outcome of AEs will be followed up and recorded. All Adverse Events (AEs) occurring during clinical studies will be recorded in the eCRF. During the study, complete reports of all AEs will be entered in the Participants site source documents, and if applicable, on the appropriate study case report forms (CRFs). A licensed clinician will be responsible for: identifying and evaluating the severity (mild, moderate, or severe) and clinical importance of the AE, taking appropriate medical action(s), and for notifying the Sponsor immediately of an SAE as specified in the protocol and for notifying the Science Department for reporting to the IRB/IEC. For any laboratory abnormality, the PI or Sub-Investigator will make a judgement as to its clinical significance. The PI or Sub-Investigator will comply with applicable regulatory requirement(s) related to the reporting of SAEs to the IRB/IEC.

The Monitor(s) will review completed CRF data and will compare CRF entries with information recorded in the source documents. Any discrepancies or omissions in either data source will be discussed with the site personnel who should make the appropriate corrections to the documents.

ELIGIBILITY:
Inclusion Criteria:

* Be able to give written informed consent.
* Be between 18-55 years of age.
* Has a BMI between >18.5 and <32.0 kg/m2.
* Has a stable body weight (≤5 % change) over the past 3-months.
* Is in general good health, as determined by the investigator.
* Consuming a single daily portion of red/processed meat in their Western diet as assessed by Food Frequency Questionnaire (meat items) at screening.
* Willing to avoid lifestyle fluctuations (diet, exercise) for the duration of the study.

Exclusion Criteria:

* Participants who are pregnant or wish to become pregnant during the study.
* Participants who are lactating and/or currently breastfeeding.
* Participants currently of biological childbearing potential, but not using a continuous effective method of contraception.
* Is hypersensitive to any of the components of the Study Product.
* Participants who have taken oral antibiotics 12 weeks prior to visit 1.
* Have a significant acute or chronic coexisting illness such as uncontrolled hypertension, uncontrolled hyperlipidaemia, hypercoagulation, inflammatory disorders, or any condition which contraindicates, in the investigator's judgement, entry to the study.
* Metabolic or chronic diseases (including pre-diabetes and diabetes), metabolic syndrome, obesity (Class 2), uncontrolled high blood pressure or chronic inflammation or any ongoing medical condition that interferes significantly with absorption and digestion and/or gastrointestinal (GI) function.
* Participants has acute or chronic gastrointestinal and/or infective disease (i.e., coeliac disease, diarrhoea, Crohn's disease, ulcerative colitis, irritable bowel syndrome, diverticulosis, stomach or duodenal ulcers, hepatitis, etc.), or with a history of such diseases or gastrointestinal surgery (appendectomy in the last 3 months acceptable).
* Has a malignant disease or any concomitant end-stage organ disease, and are severely immunocompromised (HIV positive, transplant patient, on antirejection medications, or chemotherapy or radiotherapy which, in the Investigator's judgment, contraindicates participation in the study.
* Participant has a history of drug and/or alcohol abuse at the time of enrolment (Drinks more than nationally recommended units per week (>11 units for women; >17 units for men); alcohol/substance abuse disorder).
* Is a smoker/vaper/consumes or uses nicotine containing products.
* Taking medications/supplements that the investigator believes would interfere with the objectives of the study. Prohibited medications include:
* Metformin
* Proton pump inhibitors
* Protein supplements
* Creatinine supplements
* Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the study.
* Participants may not be receiving treatment involving experimental drugs/supplements. If the Participant has been in a recent experimental study, these must have been completed not less than 60 days prior to this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2024-10-11 (Estimated); Study Completion 2024-10-18 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of replacing animal protein in a typical Western diet with plant-derived protein delivered in a (soy-based) tofu on gut microbiome composition. | 10 weeks
  Change from baseline (Week 0) to washout (Week 10) in gut microbiome composition as measured by shotgun metagenomics at weeks -2, 0,8 and 10.

SECONDARY OUTCOMES:
To evaluate the functional activity of the gut microbiome, and any alterations caused by the soya replacement. | 8 weeks
  Change from baseline (Week 0) to end of intervention (Week 8) in functional activity of the gut microbiome as measured by stool meta transcriptomics in a population comprising of healthy males and females.
To evaluate the metabolome of urine and faecal samples and any alterations caused by the soya replacement. | 8 weeks
  Change from baseline (Week 0) to end of intervention (Week 8) on:
  Urine metabolome (whole m/z ratio spectrum) Faecal metabolome (whole m/z ratio spectrum) Urine and Faecal metabolites will be measured using untargeted UHPLC-MS.
To measure the effect of the meat substitution on a panel of proinflammatory cytokines, based on the observation that particular taxa are associated with an inflammatory phenotype. | 8 weeks
  Change from baseline (Week 0) to end of intervention (Week 8) to measure the effect of the meat substitution on serum levels of the following inflammatory cytokines: TNF-alpha, IFN-alpha2, IL1b, IL3, IL4, IL6, IL7,IL8, IL22, CRP, CX3CL1 and Saa3 using MSD multiplex kits.
To measure the effect of the meat substitution on cholesterol and serum triglycerides. | 8 weeks
  Change from baseline (Week 0) to end of intervention (Week 8) on lipid profile:
  * Total cholesterol
  * Triglycerides
To measure the effect of the meat substitution on blood pressure. | 8 weeks
  Change from baseline (Week 0) to end of intervention (Week 8) on blood pressure [systolic/diastolic blood pressure (mmHg)].
To measure the effect of the meat substitution on body mass index (BMI). | 8 weeks
  Change from baseline (Week 0) to end of intervention (Week 8) on body mass index.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Dinan, Principal Investigator — Atlantia Clinical Trials; Paul W O'Toole, Study Director — University College Cork
Locations (1):
- Atlantia Clinical Trials, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No